CLINICAL TRIAL: NCT04203251
Title: Evaluation of TTE Utilization in Medical Surgery Step-Down Unit: Use of AI Assisted Point-of-Care Echo With Guidance Technology
Brief Title: Evaluation of TTE Utilization in Medical Surgery Step-Down Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Caption Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUCSF01
Record Dates: First submitted 2019-12-05; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Cardiac Disease
Keywords: Artificial Intelligence; Cardiac Monitoring
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Caption Health Guidance Technology

SUMMARY:
This is a non-randomized, un-blinded study to evaluate Caption Health guidance software in patients in the medical surgery step-down unit. Patients will be scanned by a trained hospitalist and up to 4 standard views will be obtained per participant: PLAX, PSAX-PM, AP4 and SubC4. Observations will be made regarding human factors and performance of the device.

ELIGIBILITY:
Inclusion Criteria: .

* Patients ≥18 years old
* Patients in the medical surgery step-down clinical setting
* Patients who consent to participating in the study

Exclusion Criteria: .

* ● Patients with emergent or urgent episodes of injury and illness that can lead to death or disability without rapid intervention

  * Unable to lie flat for study
  * Patients experiencing a known or suspected acute cardiac event at the time of evaluation
  * Patients with severe chest wall abnormalities
  * Patients who have undergone pneumonectomy
  * Patients with recent abdominal surgery
  * Patients unwilling or unable to give written informed consent
  * Principal Investigator determination to exclude the subject from participation
  * Investigators also have the right to withdraw patient from the study in the event of illness, adverse events, or other reasons concerning the health or well-being of the patient, or in the case of non-compliance.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in the medical surgery step down unit at UCSF.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Mean time to acquire images | Up to 3 months
  Assess the time to acquire cardiac ultrasound images with and without Caption AI Gudiance
Percentage of attempted studies with clinically useful images | Up to 3 Months
  Compare the percentage of clinically useful versus not useful images

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No